CLINICAL TRIAL: NCT04780321
Title: A Randomized, Double-blind, Placebo-controlled, Phase Ib/II Clinical Study to Evaluate the Preliminary Efficacy, Safety, Pharmacokinetic Profiles and Immunogenicity of JS016 in Participants With Mild and Moderate COVID-19 or of SARS-CoV-2 Asymptomatic Infection
Brief Title: JS016 (Anti-SARS-CoV-2 Monoclonal Antibody)With Mild and Moderate COVID-19 or SARS-CoV-2 Asymptomatic Infection Subects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS016-002-Ib/II
Record Dates: First submitted 2020-09-23; First posted 2021-03-03 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-SARS-CoV-2 Monoclonal Antibody dose 1/2/3 (Active Comparator): use Anti-SARS-CoV-2 Monoclonal Antibody,dose 1/2/3 to treat COVID-19
  Interventions: Biological: Recombinant Human Anti-SARS-CoV-2 Monoclonal Antibody(25mg/kg;50mg/kg;100mg/kg)
- Placebo (Placebo Comparator): use placebo to treat COVID-19
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Recombinant Human Anti-SARS-CoV-2 Monoclonal Antibody(25mg/kg;50mg/kg;100mg/kg) — use dose 1/2/3 60 patients receipt JS016 intravenous infusion on day 1
  Arms: Anti-SARS-CoV-2 Monoclonal Antibody dose 1/2/3
Drug: Placebo — 30 patients receipt placebo intravenous infusion on day 1
  Arms: Placebo

SUMMARY:
JS016-002-Ib/II is a randomized, double-blinded, placebo-controlled study, to investigate the safety, PK profiles, preliminary efficacy and immunogenicity of intravenous Recombinant Human Anti-SARS-CoV-2 Monoclonal Antibody (JS016) in participants with mild and moderate COVID-19 or of SARS-CoV-2 Asymptomatic Infection.

Three doses of JS016 are to be investigated, including 25mg/kg, 50mg/kg and 100mg/kg, given as single dose of intravenous infusion. In total, 90 participants will be enrolled with 30 participants each for 25, 50 and 100mg/kg dose cohort at a ratio of 2:1 to receive investigational product or placebo treatment, respectively.

DETAILED DESCRIPTION:
"Each participant will receive JS016 or matched placebo intravenous infusion on D1 (randomizing day). Non-pharmaceutical supportive background therapy (e.g. oxygen inhalation) for COVID-19 is allowed per clinical needs.

Investigators will be kept blinded to review the preliminary efficacy and safety data on a regular basis. Meanwhile, a study evaluation team (SET) composed of medical monitors, safety assessors and statisticians will be set up to review the study status, safety and preliminary efficacy of the participants at the pre-specified time points or as necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-65 years (inclusive) ,women or man
2. SARS-CoV-2 detected in the diagnostic specimen (nasopharyngeal swab)
3. High homology of viral gene sequencing with the known SARS-CoV-2."
4. Mild/moderateillness COVID-19 or SARS-CoV-2 asymptomatic infection
5. Within 7 days from the onset time of symptoms to randomization or within 5 days from the first time of SARS-CoV-2 positive test to randomization with required viral load
6. No plan of pregnancy and being willing to use effective contraceptive measures
7. Signed the informed consent form, sufficiently understanding of the content

Exclusion Criteria:

1. positive IgM/IgG against SARS-CoV-2 prior to randomization.
2. Severeor critical illness
3. Uncontrolled hypertension, cardiovascular/cerebrovascular diseases,lung diseases
4. Type 1 diabetes, or newly diagnosed or poorly controlled type 2 diabetes
5. Liver and kidney dysfunction, immune or inflammatory diseases, infections, surgery, tumors, and other major diseases
6. History of SARS-CoV-2 vaccination or participation in clinical trial with neutralizing antibody against SARS-CoV-2.
7. Use of therapeutic biologics within 3 months prior to screening, or within the elimination period (5 half-lives) of such drugs as the day of dosing
8. Has participated in any other interventional clinical study involving anstudy drug within 3 months prior to screening, or within the elimination period (5 half-lives) of the study drug as the day of dosing
9. Platelets and hemoglobin test results during screening period are abnormal and have clinical significanc.
10. Anaphylaxis, urine drug screening, alcohol dependence, lactation during pregnancy, blood loss, and others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy Measurs(Time to negative conversion in viral nucleic acid test(by RT-PCR) for diagnostic samples) | 0-85days
  Time to negative conversion in viral nucleic acid test (by RT-PCR) for diagnostic samples, negative conversion is defined as two consecutive negative nucleic acid test for diagnostic samples after randomization
Safety Measurements : 90 of participants with treatment-related adverse events as assessed byCTCAE v5.0 | 0-85days
  Any adverse event, serious adverse events (SAEs) occurring during the clinical study, including clinical symptoms and abnormal vital signs, abnormal laboratory tests (complete blood cell count, serum chemistry, routine urinalysis, coagulation function, myocardial enzymogram, etc.) and abnormality of 12-lead ECGs will be observed for all the participants

SECONDARY OUTCOMES:
PK Measures:AUC0-tau | Day 0 to Day 85
  Area under the plasma drug concentration-time curve from time 0 to one dosing interval (AUC0-tau)
PK Measures：Cmax | Day 0 to Day 85
  Maximum plasma drug concentration after administration (Cmax)
PK Measures：Tmax | Day 0 to Day 85
  Time to the maximum plasma drug concentrations after administration (Tmax)
PK Measures：t1/2 | Day 0 to Day 85
  Terminal half life (t1/2)
PK Measures：CL | Day 0 to Day 85
  Total clearance (CL)
PK Measures：Vd | Day 0 to Day 85
  Apparent volume of distribution (Vd)
Proportions of participants with negative conversion in viral nucleic acid test | Day 0 to Day 85
  Proportions of participants with negative conversion in viral nucleic acid test 7 days and 14 days after administration (performed on each day of the first week after dosing, every other day of the 2nd week, once a week from the 3rd week)
Viral load change from baseline | Day 0 to Day 85
  Viral load change from baseline (performed on each day of the first week after dosing, every other day of the 2nd week, once a week from the 3rd week)
Pulmonary CT（observe by imaging reports to degree of pulmonary inflammation, degree of vitreous fibrosis) | Day 0 to Day 85
  Pulmonary CT changes during the study period

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Ditan Hospital affiliated to Capital Medical University, Beijing
  - Huashan Hospital affiliated to Fudan University, Shanghai

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343